CLINICAL TRIAL: NCT00253513
Title: A Study of a Reduced-Intensity Conditioning Regimen With Treosulfan and Fludarabine for Allogeneic Hematopoietic Cell Transplantation for Patients With Acute Leukemia
Brief Title: Treosulfan and Fludarabine in Treating Younger Patients Who Are Undergoing a Donor Stem Cell Transplant for Acute Myeloid Leukemia, Acute Lymphoblastic Leukemia, or Myelodysplastic Syndrome
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: medac GmbH (Industry); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000445306; FHCRC-1931.00; MEDAC-FHCRC-1931.00; OHSU-HEM-05107-LM; 1765 (Other: OHSU IRB)
Record Dates: First submitted 2005-11-11; First posted 2005-11-15 (Estimated); Results first posted 2011-02-11 (Estimated); Last update posted 2012-06-01 (Estimated); Status verified 2011-02

CONDITIONS: Leukemia; Myelodysplastic Syndromes
Keywords: adult acute lymphoblastic leukemia in remission; adult acute myeloid leukemia in remission; childhood acute lymphoblastic leukemia in remission; recurrent adult acute lymphoblastic leukemia; recurrent adult acute myeloid leukemia; recurrent childhood acute lymphoblastic leukemia; recurrent childhood acute myeloid leukemia; secondary acute myeloid leukemia; myelodysplastic syndromes; childhood myelodysplastic syndromes
MeSH Terms: conditions — Leukemia; Myelodysplastic Syndromes; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute | interventions — fludarabine; treosulfan; Bone Marrow Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: fludarabine — 30 mg/m2, IV for 5 days
Drug: treosulfan — 12 or 14 g/m2, IV for 5 days
Procedure: allogeneic blood or bone marrow transplantation — bone marrow or peripheral blood stem cells

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as treosulfan and fludarabine, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Giving treosulfan and fludarabine together with a donor bone marrow transplant or a peripheral stem cell transplant may be an effective treatment for acute myeloid leukemia, acute lymphoblastic leukemia, or myelodysplastic syndrome.

PURPOSE: This phase II trial is studying giving treosulfan together with fludarabine to see how well it works in treating patients who are undergoing a donor stem cell transplant for acute myeloid leukemia, acute lymphoblastic leukemia, or myelodysplastic syndrome.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary Phase

* Determine the best dose of treosulfan when administered with fludarabine as a reduced-intensity conditioning regimen followed by allogeneic hematopoietic stem cell transplantation, in terms of incidence of severe to fatal toxicity to major organ systems and incidence of graft failure, in patients with acute myeloid leukemia, lymphoblastic leukemia, or myelodysplastic syndrome.

Secondary Phase

* Determine the safety of this regimen, in terms of incidence of grade II-IV acute and chronic graft-versus-host disease, in these patients.
* Determine, preliminarily, the efficacy of this regimen, in terms of incidence of relapse, overall and disease-free survival, donor chimerism on days 28 and 100, and incidence of 200-day and 1-year nonrelapse mortality, in these patients.
* Determine the pharmacokinetic and pharmacodynamic profile of treosulfan in patients treated with this regimen.

OUTLINE: This is a multicenter, dose-finding study of treosulfan.

* Reduced-intensity conditioning: Patients receive treosulfan IV over 2 hours on days -6 to -4 and fludarabine IV over 30 minutes on days -6 to -2.

Cohorts of 5-10 patients receive escalating/de-escalating doses of treosulfan until the best dose is determined among the 3 pre-selected doses. The best dose is defined as the dose preceding that at which 4 of 10 patients experience dose-limiting toxicity.

* Allogeneic hematopoietic cell transplantation (AHCT): Patients undergo allogeneic bone marrow or peripheral blood stem cell transplantation on day 0.

All male patients with acute lymphoblastic leukemia OR male patients with acute myeloid leukemia who have prior or current testicular involvement receive external-beam radiotherapy to the testicles before AHCT.

After completion of study treatment, patents are followed periodically.

PROJECTED ACCRUAL: A total of 60 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of acute myeloid leukemia, lymphoblastic leukemia, or myelodysplastic syndrome

  * Any phase allowed, including any of the following:

    * Disease in remission
    * Relapsed or primary refractory disease
* No CNS leukemic involvement not clearing with prior intrathecal chemotherapy and/or cranial radiotherapy
* Planning to undergo unmanipulated allogeneic bone marrow or peripheral blood stem cell transplantation

  * Filgrastim (G-CSF) mobilization of bone marrow or stem cells allowed
* Donor available, meeting 1 of the following criteria:

  * HLA-identical related donor
  * HLA-A, -B, -C, -DRB1, and -DQB1 matched unrelated donor by high-resolution DNA typing

    * A single allele mismatch allowed

PATIENT CHARACTERISTICS:

Performance status

* Karnofsky 70-100% OR
* Lansky 70-100%

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* Bilirubin ≤ 2 times upper limit of normal (ULN)
* AST ≤ 2 times ULN
* No evidence of synthetic dysfunction
* No severe cirrhosis
* No active infectious hepatitis

Renal

* Creatinine clearance ≥ 50%
* Creatinine ≤ 2 times ULN
* Dialysis independent

Cardiovascular

* No cardiac insufficiency requiring treatment
* No symptomatic coronary artery disease
* Ejection fraction ≥ 35% (for patients with history of cardiac disease or anthracycline exposure)

Pulmonary

* PO_2 ≥ 70 mm Hg AND DLCO ≥ 70% of predicted OR
* PO_2 ≥ 80 mm Hg AND DLCO ≥ 60% of predicted
* Not requiring supplementary continuous oxygen

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No other disease that would severely limit life expectancy
* No HIV positivity
* No active infection requiring deferral of conditioning
* No known hypersensitivity to the study drugs

PRIOR CONCURRENT THERAPY:

Biologic therapy

* See Disease Characteristics
* No prior allogeneic bone marrow or stem cell transplantation
* No concurrent umbilical cord blood or autologous transplantation

Chemotherapy

* See Disease Characteristics

Radiotherapy

* See Disease Characteristics

Other

* More than 4 weeks since prior experimental drugs
* Concurrent enrollment on another protocol for graft-versus-host disease prophylaxis allowed

Max Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2005-06; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eneida Nemecek, MD, Principal Investigator — OHSU Knight Cancer Institute
Locations (3):
- United States (3):
  - OHSU Knight Cancer Institute, Portland, Oregon
  - Seattle Cancer Care Alliance, Seattle, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients recruited at OHSU Knight Cancer Institute clinics in Portland, Oregon and Fred Hutchinson Cancer Research Center or University of Washington Medical Center clinics, Seattle, Washington.
Groups:
- Treosulfan and Fludarabine Conditioning: Conditioning with Treosulfan (12 or 14 g/m2, IV for 5 days) and Fludarabine (30 mg/m2, IV for 5 days) followed by Allogeneic Hematopoietic Cell Transplantation for High-Risk Hematologic Malignancies
Period: Overall Study
Arm/Group | Treosulfan and Fludarabine Conditioning
Started | 60
Completed | 60
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treosulfan and Fludarabine Conditioning
Number analyzed (Participants) | 60
Age, Customized [Number; unit: Participants]
  < 21 years | 10
  Between 21 - 50 years | 31
  Between 50 - 60 years | 19
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36
  Male | 24
Region of Enrollment [Number; unit: participants]
  United States | 60
Disease status at transplantation [Number; unit: Participants]
  Acute Lymphoblastic Leukemia(ALL)2nd/3rd remission | 3
  Acute Myelogenous Leukemia(AML)1st remission | 26
  AML, 2nd or greater remission. | 10
  AML, relapsed or primary refractory | 8
  Myelodysplastic Syndrome(MDS): Refract. Anemia(RA) | 6
  MDS: RA with excess blasts in transformation | 7
Disease risk group [Number; unit: Participants] — Low-risk disease: AML or ALL in first remission, MDS with IPSS (International Prognosis Scoring System)=0; standard risk: ALL or AML in second or greater remission, MDS with IPSS 0.5-2; high risk: relapsed/refractory ALL or AML, MDS with IPSS>=2.5.
  Participants
    Low - AML/ALL in 1st rem., MDS with IPSS=0 | 26
    Standard (ALL or AML in 2nd or greater rem.) | 22
    High -relapsed/refract. ALL/AML/MDS w/ IPSS>=2.5 | 12
Cytogenetic risk group [Number; unit: Participants] — Good risk cytogenetics: t(8;21), t(15;17), or inversion 16 for AML, hyperdiploidy for ALL, -Y, del(5q), del(20q), or normal for MDS; poor risk: 11q23 abnormalities, monosomy 7, monosomy 5, deletion 5q, or abnormalities of 3q for AML, t(9;22) or extreme hypodiploidy for ALL, chromosome 7 abnormalities in MDS,$3 chromosome abnormalities for any disease type; Intermediate risk: all others
  Participants
    Good | 16
    Intermediate | 8
    Poor | 36
Hematopoietic Cell Transplantation Comorbidity Index (HCT CI) [Number; unit: Participants] — Risk of mortality after allograft (0 is lower risk, >=3 is higher risk)
  Participants
    0 | 13
    1-2 | 19
    >=3 | 28
Donor type [Number; unit: participants]
  HLA (human leukocyte antigen) -identical sibling | 30
  HLA-matched unrelated donor | 30
Stem cell source [Number; unit: participants]
  Bone marrow | 7
  Filgrastim-mobilized PBPC | 53

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Experiencing Regimen-related Toxicity Events in Study Population
Description: Proportion of patients experiencing regimen-related toxicity to major organ systems from day minus 6 to day 28. Major organ systems: cardiac, bladder/renal, pulmonary, hepatic, neurologic and gastrointestinal
Time Frame: 34 days and 2 years
Measure: Number; unit: participants
Arm/Group | Treosulfan and Fludarabine Conditioning
Number analyzed (Participants) | 60
participants
  Severe Regimen Related Toxicity (RRT) | 2
  Nonrelapse mortality at 2 years | 5

2. Primary Outcome: Number of Patients Experiencing Graft Failure
Description: Graft versus Host Disease (GVHD) is a frequent complication of allogeneic bone marrow transplant in which the engrafted donor cells attacks the patient's organs and tissue. Acute GVHD (aGVHD) usually occurs during the first three months following an allogeneic BMT. Chronic GVHD (cGVHD) usually develops after the third month post-transplant. Patients may experience one, both or neither.
Time Frame: 42 days
Population: For graft failure 2 of the 60 patients were not evaluable because they exeperienced another event (relapsed) before they could be evaluable for graft failure.
Measure: Number; unit: participants
Arm/Group | Treosulfan and Fludarabine Conditioning
Number analyzed (Participants) | 58
participants
  acute graft vs. host disease (aGVHD) | 36
  chronic graft vs. host disease (cGVHD) | 31

3. Primary Outcome: Incidence (Percent of Participants) With Nonrelapse Mortality (NRM) by Day 200 (Secondary Phase Only)
Description: NRM (Non relapse mortality) - death not attributed to the primary cancer.
Time Frame: 200 days
Measure: Number (95% Confidence Interval); unit: percent of participants
Arm/Group | Treosulfan and Fludarabine Conditioning
Number analyzed (Participants) | 60
percent of participants | 5 [0 to 10.5]

4. Secondary Outcome: Number of Subjects Who Are Without Disease at One Year as Indicator of Disease Free Survival.
Time Frame: One year
Measure: Number; unit: participants
Arm/Group | Treosulfan and Fludarabine Conditioning
Number analyzed (Participants) | 60
participants | 58

ADVERSE EVENTS:
Arm/Group | Treosulfan and Fludarabine Conditioning
Serious Adverse Events (participants affected / at risk) | 5/60
Other Adverse Events (participants affected / at risk) | 0/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treosulfan and Fludarabine Conditioning (N=60)
Grade 4 mucositis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Death - cGVHD (Immune system disorders) | 2 (2)
Death - intracranial hemmorrage (Blood and lymphatic system disorders) | 1 (1)
Death - fungal infection (Infections and infestations) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No